CLINICAL TRIAL: NCT00217633
Title: Prospective Evaluation of Pelvic Exenteration in Patients With Recurrent Cervical Cancer
Brief Title: Pelvic Exenteration in Treating Patients With Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0222; NCI-2009-00593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000442396; GOG-0222 (Other: Gynecologic Oncology Group); GOG-0222 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

ARMS (1):
- Treatment (pelvic exenteration) (Experimental): Patients undergo pelvic exenteration within 14 days after study entry.
  Interventions: Procedure: Conventional Surgery

INTERVENTIONS:
Procedure: Conventional Surgery

SUMMARY:
This phase II trial is studying how well pelvic exenteration works in treating patients with recurrent cervical cancer. Pelvic exenteration may be effective in treating recurrent cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Correlate progression-free survival and overall survival with tumor size, time interval between primary cancer management and pelvic exenteration, and presence or absence of pelvic sidewall fixation by clinical examination in patients with recurrent cervical cancer treated with pelvic exenteration.

SECONDARY OBJECTIVES:

I. Determine quality of life of patients treated with this procedure. II. Correlate quality of life with reconstructive technique (e.g., no ostomy or ≥ 1 ostomy) in patients treated with this procedure.

OUTLINE:

Patients undergo pelvic exenteration within 14 days after study entry. Quality of life is assessed at baseline and at 6, 12, and 24 months after surgery. After completion of study treatment, patients are followed within 30 days, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical cancer

  * Any histology
  * Documented or suspected central pelvic disease with or without pelvic sidewall fixation from tumor and/or radiation fibrosis
* Meets 1 of the following stage criteria:

  * Recurrent disease, defined as reappearance of disease after a complete clinical response lasting ≥ 1 month
  * Persistent disease, defined as presence of disease by biopsy ≥ 3 months after completion of primary therapy
* Must have received prior primary treatment, including any of the following:

  * Surgery with or without post operative radiotherapy with or without chemotherapy
  * Primary radiotherapy with or without chemotherapy
  * Neoadjuvant chemotherapy followed by surgery
  * Neoadjuvant chemotherapy followed by surgery with or without radiotherapy or chemotherapy
* Plans to undergo pelvic exenteration to remove the pelvic disease within 14 days after study entry

  * Deemed to be a good surgical candidate

    * No evidence of distant disease or disease that is felt to be unresectable by physical examination
    * Patients with suspicious pelvic or para-aortic nodal disease as the only site(s) of extrapelvic disease are eligible at the discretion of the surgeon
  * Patients whose surgery is planned solely for managing complications (e.g., rectovaginal fistula, vesicovaginal fistula) of disease or prior therapy are not eligible
  * Patients whose surgery is planned as a prophylactic measure due to a slow or suboptimal clinical or radiographical tumor response during the course of primary therapy are not eligible
* No distant site of metastases by CT scan or MRI of the abdomen/pelvis OR positron-emission tomography
* No noncervical primary tumor
* No prior anterior or posterior pelvic exenteration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From entry to protocol to death; or for living patients, the date of last contact, up to 93 years
Progression-free survival | From study entry to date of reappearance or increasing parameters of disease or death, or to date of last contact for patients without disease progression, up to 93 years

SECONDARY OUTCOMES:
Impact of surgery therapy (exenteration and reconstructive surgery type) on quality of life assessed by Functional Assessment of Cancer Therapy-Cervix (FACT-CX) | At baseline, 6, 12, and 24 months post exenteration

CONTACTS AND LOCATIONS:
Overall Officials: D. McMeekin, Principal Investigator — Gynecologic Oncology Group
Locations (39):
- United States (38):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Gynecologic Oncology Group, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Auburn Regional Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
- M D Anderson International Spain, Madrid, Madrid, Spain